CLINICAL TRIAL: NCT02094196
Title: The Role of Dopaminergic and Glutamatergic Neurotransmission for Dysfunctional Learning in Alcohol Use Disorders (LeAD P5)
Brief Title: The Role of Dopaminergic and Glutamatergic Neurotransmission for Dysfunctional Learning in Alcohol Use Disorders
Acronym: LeADP5
Status: Completed | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Collaborators: Charite University, Berlin, Germany (Other)
Responsible Party: Sponsor
Other Study IDs: GA707/6-1
Record Dates: First submitted 2014-03-20; First posted 2014-03-21 (Estimated); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Alcohol Use Disorder
Keywords: Reward- based learning; Pavlovian-to-instrumental transfer; Relapse Risk; Positron emission tomography (PET); Magnetic resonance spectroscopy (MRS); Dopamine receptor availability; Glutamate
MeSH Terms: conditions — Alcoholism | interventions — Ethanol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Bloodsample are taken for genetic analysis
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Controls, highrisk for AD: Community-based ad-hoc participants, high risk for alcohol dependence, matched to inpatients by sociodemographics
- Controls, low risk for AD: Community-based ad-hoc participants, low risk for alcohol dependence, matched to inpatients by sociodemographics
- Alcohol detoxification: Inpatients with alcohol dependence from local psychiatric hospital wards (18-65 years old)
  Interventions: Other: Alcohol detoxification

INTERVENTIONS:
Other: Alcohol detoxification — Detoxified alcohol- dependent patients in an inpatient setting
  Other Names: Alcohol- dependent patients
  Groups: Alcohol detoxification

SUMMARY:
The aim of this project is to assess reward- based learning behavior and its association with alterations in dopaminergic and glutamatergic transmission in detoxified alcohol-dependent patients and matched controls.

The investigators will explore how these alterations interact with clinical and psychosocial factors which can modify the relapse risk and learning deficits.

Patients will be detoxified in an inpatient setting. Clinical assessments, behavioral paradigms of learning and brain imaging will be carried out within at least 4 half- lives after any psychotropic medication.

The investigators will implement and apply functional imaging paradigms assessing Pavlovian-to-instrumental transfer and reversal learning tasks and associate model parameters of learning with alcohol craving, intake and prospective relapse risk.

In this project, the impact of the dopamine x glutamate interaction on learning deficits and consecutive relapse probability is targeted with [18F]fallypride PET and the measurement of absolute concentrations of glutamate with magnetic resonance spectroscopy (MRS).

DETAILED DESCRIPTION:
Alcohol consumption despite negative consequences may rely on impaired flexibility in adapting the behavior to environmental changes, i.e. learning in response to reward contingencies. This learning deficit is of clinical relevance particularly during therapy and for the psychosocial outcome.

The reduced availability of central dopamine D2-receptors in detoxified alcohol dependent patients observed in PET investigations and their hypothetical effects on reward-related learning are in line with evidence for learning deficits in hypodopaminergic states, particularly for avoidance learning in non-dependent samples. Growing evidence indicates that the learning-related striatal dopamine signals are modulated by higher executive functions involving, e.g., the prefrontal cortex.

Here, broad glutamatergic outputs of the prefrontal cortex are crucial for subcortical learning mechanisms and match with recent models of interactive dopamine-glutamate dysfunctions and models of neurotrophic signaling in alcohol dependence.

ELIGIBILITY:
Inclusion Criteria:

* Alcohol dependence according to DSM-IV
* Minimum of 72 hours of abstinence, maximum of 21 days of abstinence
* Minimum of three years of alcohol dependence
* Low severity of withdrawal symptoms
* Ability to provide fully informed consent and to use self- rating scales

Exclusion Criteria:

* Lifetime history of DSM- IV bipolar or psychotic disorder
* Current threshold DSM-IV diagnosis of any following disorders: current major - depressive disorder, generalized anxiety disorder, PTSD, borderline personality disorder or obsessive- compulsive disorder
* History of substance dependence other than alcohol or nicotine dependence

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Detoxified alcohol- dependent patients and age- and gender matched healthy controls living in Germany
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Striatal D2-receptor availability (PET) and prefrontal glutamate concentration (MRS) | first assessment time point (alc. dependent pat. up to 21 days after detoxification)
  reduction in striatal D2-receptor availability and a increase in prefrontal glutamate concentration in alcohol-dependent patients compared to healthy controls

SECONDARY OUTCOMES:
behavioral data in reward-habit-learning paradigms | first assessment time point (alc. dependent pat. up to 21 days after detoxification)
  Reduced learning speed and PIT withdrawal score in the probabilistic reversal learning task
Treatment response | 12-month follow-up period beginning after first assessment timepoint
  test the predictive effects of striatal D2-receptor availability and prefrontal glutamate availability for treatment outcome (relapse vs abstinence) in alcohol-dependent patients

OTHER OUTCOMES:
striatal-prefrontal connectivity (fMRI) | first assessment time point (alc. dependent pat. up to 21 days after detoxification)
  striatal-prefrontal connectivity (see other LeAD-projects) in the probabilistic reversal learning task

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Gallinat, Prof MD, Principal Investigator — Charite University, Berlin, Germany; Andreas Heinz, Prof MD, Study Chair — Charite University, Berlin, Germany; Hans-Ulrich Wittchen, Prof PhD, Study Director — Technische Universität Dresden, Dresden, Germany
Locations (2):
- Germany (2):
  - Charité Berlin, Division of Neuroimaging, Berlin
  - Charité - Universitätsmedizin Berlin, Berlin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Spitta G, Gleich T, Maricic LM, Rosenthal A, Schubert F, Aydin S, Heinz A, Gallinat J. Reduced GABA Levels in the ACC of Actively Drinking High Risk Individuals Compared to Recently Detoxified Alcohol-Dependent Patients. J Integr Neurosci. 2024 Oct 14;23(10):190. doi: 10.31083/j.jin2310190. PMID 39473159
- See also: English study description — http://gepris.dfg.de/gepris/projekt/209293518